CLINICAL TRIAL: NCT02954783
Title: Effect of Different Exercise Regimens on Intratumoral Natural Killer (NK) Cell Variability in Men With Localized Prostate Cancer Undergoing Radical Prostatectomy - a Randomized Controlled Pilot Study
Brief Title: PROstaTe Cancer - Exercise-STudy (PRO-TEST)
Acronym: PRO-TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sissal Sigmundsdóttir Djurhuus, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: H-16034670
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Localized; Exercise; Physical activity; Natural killer cells; Immune cells
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Interval Training (Experimental): The HIIT-group will receive usual care plus a supervised aerobic High Intensity Interval Training program consisting of 4 weekly sessions of approximately 35 minutes.
  Interventions: Behavioral: High Intensity Interval Training
- Usual Care Observational Control (Active Comparator): Patients randomized to usual care control will receive the standard patient care program as provided by the Department of Urology, Rigshospitalet.
  Interventions: Behavioral: Usual Care Observational Control

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Supervised aerobic High Intensity Interval Training program consisting of 4 weekly sessions of approximately 35 minutes. Patients will perform a test of maximum cardio-respiratory (VO2 peak test). Using the patient's individual wattmax, a personalized exercise program will be prescribed.
  After a light warm-up, patients will perform 25 min of aerobic high intensity interval training on a stationary bicycle, intervals will consist of cycles of HI intervals with 120% of wattmax for 1 min followed by recovery for 3 min at 30% of wattmax. Each session will be supervised by trained instructors to ensure proper technique, and progression in training load.
  Arms: High Intensity Interval Training
Behavioral: Usual Care Observational Control — The reference group will receive the standard patient care program as provided by the Department of Urology, Rigshospitalet.This includes information regarding smoking cessation and alcohol reduction and a physiotherapist consultation regarding pelvic floor exercises. This group is allowed to exercise on their own initiative or participate in any standard care hospital- or municipality-based exercise program. This will be monitored by self-report.
  Arms: Usual Care Observational Control

SUMMARY:
Background and purpose: The purpose of this study is to investigate the effect of exercise on intratumoral natural killer (NK)-cell variability in patients with localized prostate cancer undergoing radical prostatectomy.

The primary hypothesis is that exercise induces epinephrine-mediated intratumoral natural killer (NK)-cell infiltration in patients with localized prostate cancer, and that the infiltration is greater in patients performing High Intensity Interval Training compared to usual care controls.

Currently there is a lack of randomized controlled trials examining different types of exercise in patients with localized prostate cancer. Moreover there is a need for studies including biological measurements to allow a full assessment of the effect of exercise on diverse biomarkers and mechanistic pathways, which may influence cancer survival.

Subjects: Patients with histologically verified prostate adenocarcinoma scheduled for radical prostatectomy at Urologic Department, Rigshospitalet, Copenhagen, Denmark.

Methods: In this randomized controlled pilot study 30 patients with localized prostate cancer undergoing radical prostatectomy will be included and randomized 2:1 to either High Intensity Interval Training (HIIT) exercise intervention or observational control receiving usual care from inclusion and until planned surgery (radical prostatectomy).

All patients will undergo assessments at inclusion (baseline) and at follow-up after the exercise intervention period (maximum 8 weeks) 3-5 days prior to surgery.

Assessments include: anthropometrics; blood pressure; resting hearth rate; cardiorespiratory fitness by cardiopulmonary exercise test (VO2 peak.); body composition by DXA scan; quality of life by self-report questionnaires; fasting blood sample measuring cholesterol, triglycerides, insulin, c-peptide, HbA1c, glucose, hormones and inflammatory markers.

Biological tissue from tumor (primary prostate biopsies) will be retrieved from the respective local pathological departments and from the perioperative prostate specimen and sent to protocol analyses.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of exercise on the variability of intratumoral Natural Killer (NK)-cell infiltration in tumor biopsies taken before and after an exercise intervention in patients randomized 2:1 to one of two study arms: I) High Intensity Interval Training (HIIT) (N=20) or II) usual care, prior to radical prostatectomy.

In addition to this the investigators wish to investigate the effect of HIIT exercise on the infiltration of other immune cells into the tumor, tumor vessel morphology, modulation of tumor-metabolism, -biology and signaling.

Finally the aim is to explore the effect of pre-operative HIIT exercise on physiological (e.g. cardiovascular fitness, body composition, metabolic profile and metabolic inflammatory markers) and psycho-social (e.g. fatigue, emotional well-being, anxiety) endpoints relative to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified localized prostate cancer
* Eligible for curative radical prostatectomy

Exclusion Criteria:

* Any other known malignancy requiring active treatment
* Performance status > 1
* Ongoing treatment with beta blockers
* Physical disabilities precluding physical testing and/or exercise
* Inability to read and understand Danish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Variability in intratumoral Natural Killer (NK)-cell infiltration | Primary prostate biopsies and up to 8 weeks
  Natural killer (NK)-cell infiltration will be quantified using histological analyses.

SECONDARY OUTCOMES:
Tumor vessel morphology | Primary prostate biopsies and up to 8 weeks
  Tumor vessel morphology will be evaluated using histological analyses.
Tumor-metabolism, - biology and signaling | Primary prostate biopsies and up to 8 weeks
  Tumor samples will undergo proteomic analyzes in order to uncover potential upregulated biomarkers.
Changes in immune cells | Baseline and up to 8 weeks
  Quantification of immune cells will be measured in blood samples by flowcytometry analyses.
Changes in epinephrine concentration | Baseline and up to 8 weeks
  Concentrations of epinephrine will be measured in blood samples by radioimmunoassay analyses.
Changes in nor-epinephrine concentration | Baseline and up to 8 weeks
  Concentrations of nor-epinephrine will be measured in blood samples by radioimmunoassay analyses.
Changes in IL-1 concentration | Baseline and up to 8 weeks
  Concentrations of IL-1 (Interleukin 1) will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in IL- 2 concentration | Baseline and up to 8 weeks
  Concentrations of IL-2 (Interleukin 2) will be measured in fasting blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in IL- 6 concentration | Baseline and up to 8 weeks
  Concentrations of IL-6 (Interleukin 6) will be measured in fasting blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in IL- 8 concentration | Baseline and up to 8 weeks
  Concentrations of IL-8 (Interleukin 8) will be measured in fasting blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in IL- 10 concentration | Baseline and up to 8 weeks
  Concentrations of IL-10 (Interleukin 10) will be measured in fasting blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in IL- 15R alpha complex concentration | Baseline and up to 8 weeks
  Concentrations of IL- 15Rα (IL- 15 receptor alpha) complex will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in Tumor Necrosis Factor alpha (TNFa) concentration | Baseline and up to 8 weeks
  Concentrations of TNFa will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in Interferon Gamma (IFNγ) concentration | Baseline and up to 8 weeks
  Concentrations of IFNγ will be measured in blood samples by Enzyme-Linked Immunosorbent Assay (ELISA) analyses.
Changes in Plasma Total-Cholesterol concentrations | Baseline and up to 8 weeks
  Concentrations of total cholesterol will be measured in fasting blood samples by standard laboratory methods.
Changes in Plasma LDL-Cholesterol concentrations | Baseline and up to 8 weeks
  Concentrations of LDL-cholesterol will be measured in fasting blood samples by standard laboratory methods
Changes in Plasma HDL-Cholesterol concentrations | Baseline and up to 8 weeks
  Concentrations of HDL-cholesterol will be measured in fasting blood samples by standard laboratory methods
Changes in Plasma Triglyceride concentrations | Baseline to and up to 8 weeks
  Concentrations of triglycerides will be measured in fasting blood samples by standard laboratory methods
Changes in HbA1C (fasting blood samples) | Baseline and up to 8 weeks
  Concentrations of HbA1C will be measured in fasting blood samples by standard laboratory methods
Changes in insulin | Baseline and up to 8 weeks
  Concentrations of Insulin will be measured in fasting blood samples by standard laboratory methods
Change in body composition | Baseline and up to 8 weeks
  Body weight and anthropometrics (height, waist and hip circumference) will be assessed using standard procedures. Resting heart rate and blood pressure (Microlife, BPA100) will be determined in a supine position. Body composition (fat mass, bone mass and fat-free mass) and bone mineral density are analyzed by whole-body dual-energy X-ray absorptiometry (DXA) scan (Lunar, Lunar Corporation Madison, Wisconsin, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body. Since the different chemical compounds in the body absorb the intensity of the X-rays differently, the scan allows for a valid determination of bone mass, fat mass and fat-free/bone-free mass
Change in VO2peak | Baseline and up to 8 weeks
  The participants will undergo a maximal graded exercise test on a bicycle ergometer for evaluation of cardiovascular function and determination of the peak oxygen uptake (VO2peak). The test starts with a 5 min warm up at 70 watt (the watts may have to be adjusted to the individual fitness level). Warm up is immediately followed by a 20 watt increase every 1 min until exhaustion. Ventilation and expired gases will be measured during the test via an indirect calorimetric system, and heart rate will be assessed simultaneously.
Change in wattmax | Baseline and up to 8 weeks
  The participants will undergo a maximal graded exercise test on a bicycle ergometer for evaluation of cardiovascular function and determination of the maximum watt (wattmax). The test starts with a 5 min warm up at 70 watt (the watts may have to be adjusted to the individual fitness level). Warm up is immediately followed by a 20 watt increase every 1 min until exhaustion. The maximum watt will be calculated.
Changes in patient-reported Quality of Life - FACT | Baseline and up to 8 weeks
  Patient reported quality of life is measured by Functional Assessment of Cancer Treatment (FACT)
Changes in Sleep Quality | Baseline up to 8 weeks
  Patient reported sleep quality is measured by the Pittsburgh Sleep Quality Index (PSQI) questionaire.
Changes in Anxiety and Depression | Baseline up to 8 weeks
  Patient reported Anxiety and Depression is measured by the Hospital Anxiety and Depression Scale (HADS).
Changes in Physical Activity level | Baseline up to 8 weeks
  Patient reported physical activity is measured by the International Physical Activity Questionaire (IPAQ) - short form.
T-cell infiltration | Primary prostate biopsies from baseline and up to 8 weeks
  T-cell infiltration will be quantified using histological analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Djurhuus SS, Simonsen C, Toft BG, Thomsen SN, Wielsoe S, Roder MA, Hasselager T, Ostergren PB, Jakobsen H, Pedersen BK, Hojman P, Brasso K, Christensen JF. Exercise training to increase tumour natural killer-cell infiltration in men with localised prostate cancer: a randomised controlled trial. BJU Int. 2023 Jan;131(1):116-124. doi: 10.1111/bju.15842. Epub 2022 Jul 18. PMID 35753072